CLINICAL TRIAL: NCT00676962
Title: Facilitating Implementation of Cognitive Behavioral Therapy in Primary Care and Community Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael R. Kauth, PhD, Associate Director for Education, SC MIRECC, South Central VA Mental Illness Research, Education & Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H-22908
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Depression
Keywords: Implementation; facilitation; psychotherapy; training
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Facilitation (Experimental): Therapists receive assistance with adopting CBT
  Interventions: Behavioral: External facilitation

INTERVENTIONS:
Behavioral: External facilitation — Study facilitator meets regularly with therapists to aid implementation of CBT
  Other Names: Facilitation

SUMMARY:
The investigators propose to test the effect of external facilitation on the extent that brief cognitive behavioral therapy (CBT) for depression is incorporated into routine practice in primary care and community based clinics in the VA. The investigators will provide training in brief CBT to mental health providers in participating clinics. To the investigators' knowledge, this will be the first study of the effect of external facilitation on outcomes of a training intervention.

DETAILED DESCRIPTION:
We will test the effect of external facilitation on the extent that brief CBT for depression is incorporated into routine practice in primary care and community based clinics in the VA. We will provide training in brief CBT to mental health providers in participating clinics. To our knowledge, this will be the first study of the effect of external facilitation on outcomes of a training intervention.

ELIGIBILITY:
Inclusion Criteria:

* mental health clinicians in selected clinics who do or are willing to do psychotherapy.

Exclusion Criteria:

* clinicians who do not do psychotherapy in eligible clinics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
CBT progress notes | Monthly post-training for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Kauth, PhD, Principal Investigator — South Central MIRECC
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States